# Probing Participation in Soft Tissue Sarcoma Research: An Observational Study of Soft Tissue Sarcoma Clinical Trials

An Informed Consent Form For Power Clinical Trial's

Observational Study Involving Patients in Soft Tissue Sarcoma

Clinical Trials

Date: February 9, 2024

#### Introduction

This informed consent process serves as an introduction to our ongoing observational clinical study regarding individual decision-making within the context of soft tissue sarcoma clinical trials. We aim to understand factors influencing individuals' decisions to join, persist, or withdraw from such trials.

Participation is entirely voluntary, and you retain the right to withdraw at any point without repercussions. However, your informed consent is essential for your inclusion in the study.

#### Key details include:

- Study Goals: To identify factors impacting engagement in soft tissue sarcoma clinical trials, thereby informing strategies for enhanced participant recruitment and retention.
- Study Procedures: Primarily involving standardized questionnaires and follow-up phone calls, the study endeavors to minimize potential participant risks.

- Benefits: While immediate personal benefits may be limited, the collected data will ultimately benefit individuals with soft tissue sarcoma by contributing to improved clinical trial design and effectiveness.
- Confidentiality: All participant information will be handled with the utmost confidentiality, adhering to strict ethical and legal guidelines.

We encourage you to carefully review the enclosed consent form and discuss any questions with designated research personnel, healthcare providers, or trusted advisors. Your informed decision regarding participation is paramount.

Your Role in Advancing Soft Tissue Sarcoma Research

Soft Tissue Sarcoma clinical trials are essential for uncovering better treatments, but ensuring diverse participation remains a challenge. This study seeks to understand the factors that influence your decisions about joining, staying in, or rejoining these trials. Your insights are crucial for shaping future research to become more relevant and impactful.

We prioritize enrolling a diverse group of participants. We want to know how factors like age, race, income, and education affect your participation choices. By understanding these influences, we can develop more effective strategies to engage underrepresented groups in future trials.

Participating is entirely voluntary, and you can withdraw at any time without penalty. The study involves minimal risk and primarily consists of questionnaires and follow-up phone calls. Please carefully review the consent form and ask any questions you may have.

By sharing your experiences, you can help us develop more inclusive and effective clinical trials, ultimately leading to better treatments for this condition.

Your Role in Shaping Soft Tissue Sarcoma Research: Join Our Participant-Led Study

This observational study seeks your valuable insights! We aim to understand why individuals with soft tissue sarcoma choose to participate, remain in, or withdraw from

clinical trials. Your firsthand experiences are crucial for shaping future research and improving outcomes.

Whether you actively participated in a past study or are considering a current one, we welcome your participation. We leverage both volunteer outreach and electronic medical records to identify potential participants.

Your complete understanding of the study is paramount. Upon expressing interest, you receive a clear and comprehensive informed consent form outlining the study's goals and your rights. Bi-weekly surveys gather demographics, medical history, and your perspectives on clinical trial participation. Additionally, in-depth quarterly phone or video interviews offer an opportunity to share your voice in greater detail.

Our analysis will reveal the key factors influencing participation, informing future trial design, recruitment strategies, and retention efforts. By joining our study, you play a vital role in shaping the future of soft tissue sarcoma research.

Participation is entirely voluntary, and withdrawal is possible at any point without penalty. Completing surveys and participating in interviews involve minimal risk, with our readily available research team always available to address any questions or concerns.

Understanding the Benefits of Soft Tissue Sarcoma Observational Trials

Observational clinical trials offer soft tissue sarcoma patients a transparent and ethically sound platform to contribute to medical research. While participants do not receive experimental medications, they benefit from comprehensive medical care and gain valuable insights into their condition.

The decision to participate requires careful consideration. Patients are encouraged to engage in open and honest dialogue with their healthcare providers and the research team to fully understand the potential benefits and risks within the context of their individual needs and goals.

Participating in these trials allows patients to contribute valuable data that helps researchers gain a deeper understanding of soft tissue sarcoma's natural progression and the efficacy of existing treatments. This knowledge directly informs the development of more effective therapies, ultimately empowering patients to make informed decisions about their healthcare future.

Joining an observational trial empowers patients to become informed participants in their healthcare journey, contributing to improved understanding and future treatment options for themselves and others, all while safeguarding their individual rights and well-being.

Transparency and Choice: A Look at the Risks in soft Tissue Sarcoma Observational Studies

Observational studies of soft tissue sarcoma provide a valuable avenue for research while offering a non-invasive approach. However, it's crucial to acknowledge potential risks before making an informed decision about participation. These may include data privacy considerations, emotional challenges related to the study topic, and minimal risks associated with study procedures.

The research team is committed to complete transparency. The informed consent document clearly outlines all potential risks, along with the study's benefits and the comprehensive safeguards in place to protect your data and well-being.

You have the absolute right to ask questions, address any concerns, and request further clarification before deciding to participate. The research team is available to provide detailed information and ensure you fully understand the potential implications of participation.

Ultimately, the decision to participate rests solely with you. You have the autonomy to withdraw at any point without penalty. Your comfort and well-being are paramount, and the research team is dedicated to respecting your autonomy and addressing any concerns you may have throughout the study.

Understanding What Will Terminate Your Clinical Trial Involvement

Your journey in a clinical trial can be invaluable for medical progress, but it's essential to remember that premature endings are sometimes unavoidable. Researchers or sponsors might need to conclude the trial early due to unforeseen circumstances like funding limitations, safety concerns, or a shift in research priorities.

Furthermore, individual factors like changes in your health, unexpected pregnancy, new information prompting reevaluation, or challenges adhering to study protocols may also lead to early termination. Careful consideration and open communication about these

possibilities before enrolment are crucial for shared responsibility and informed participation.

Both you and the research team share a responsibility to ensure a beneficial and safe research experience. The informed consent document provides transparent details about potential early termination scenarios, alongside your rights and responsibilities as a participant. Additionally, the research team is committed to open communication and addressing any questions or concerns you may have throughout the trial.

Remember, even if the journey ends sooner than anticipated, your contributions and experiences hold value. You retain the right to withdraw at any time, with or without reason, and without penalty. The research team prioritizes respectful communication and strives to address any concerns you may have throughout the process.

#### A Look at Soft Tissue Sarcoma Research Opportunities

Participation in clinical studies investigating soft tissue sarcoma is entirely voluntary, and you retain the autonomy to withdraw at any stage without penalty.

Gain insights into the global <u>soft tissue sarcoma research</u> landscape by visiting Clinicaltrials.gov, a valuable resource managed by the National Institutes of Health (NIH). This platform hosts information on numerous active studies across the globe, enabling you to customize your search based on your specific location and medical concerns.

Moreover, Power's reference page offers a current listing of ongoing <u>soft tissue sarcoma</u> <u>clinical trials</u> actively seeking participants. Utilize these resources to engage collaboratively in the research process and discover options that align with your values and objectives.

Remember, your decision impacts not only your well-being but also the advancement of scientific knowledge. Carefully consider the available information, seek guidance from healthcare professionals, and choose the path that allows you to contribute meaningfully to the fight against soft tissue sarcoma.

Explore Online Resources on Diversity in Clinical Trials

As individuals seeking comprehensive information on clinical trial diversity, understanding the landscape is essential. This online world offers valuable resources to guide your decisions:

Baxter, Sally L. "Representation matters—diversity in retina clinical trials." *JAMA ophthalmology* 140, no. 11 (2022): 1103-1104.

Herremans, Kelly M., Andrea N. Riner, Robert A. Winn, and Jose G. Trevino. "Diversity and inclusion in pancreatic cancer clinical trials." *Gastroenterology* 161, no. 6 (2021): 1741-1746.

By exploring these resources, you gain the insights needed to make informed decisions about clinical trial participation. Remember, your informed choices can contribute to fostering greater inclusivity in research, ultimately benefiting both individuals and the scientific community.

### Data Privacy and Your Role in This Research

You play a vital role in this research, and protecting your privacy is paramount. While absolute confidentiality is not always possible, we have implemented robust measures to safeguard your data. It's important to understand that legal requirements may necessitate the disclosure of personal information in certain situations.

However, we prioritize your anonymity in all research publications and presentations by omitting your name and any other personally identifiable details.

Some entities, like accrediting bodies, government agencies (FDA, OHRP), safety monitors, study sponsors, and authorized representatives, may access your medical information for specific purposes related to research, quality assurance, and data analysis.

In some cases, we may request your "Authorization Form" outlining how your information will be used and shared within this study. Your explicit consent will always be sought before sharing your information or research samples with Power researchers, other institutions, or external commercial entities for future research endeavors. Remember, your confidential data will be handled securely and disposed of appropriately when no longer needed.

By understanding your rights and participating actively in decision-making regarding your data, you contribute to a research environment that prioritizes both scientific advancement and individual privacy.

## **Understanding Your Consent Rights**

Signing this consent form signifies your understanding and agreement to the following terms, ensuring your rights as a participant are protected:

- You have independently reviewed and compounded the entirety of this informed consent form, with the freedom to explore diverse perspectives before making a decision.
- We have addressed all your questions regarding the research project and its methods to your satisfaction, empowering you to participate with complete understanding.
- You have actively engaged in considering the potential benefits, drawbacks, and alternative options associated with your involvement in the research.
- Your voluntary participation in this study does not compromise your legal rights in any way.
- We are committed to keeping you informed and promptly communicating any significant updates that could impact your decision to continue participating in the research.
- Signing this consent form allows you to voice any final questions or concerns before confirming your participation.

By understanding these key points, you retain control over your decision and participate in the research on your own terms.

| Participant's Signature | | |
|-------------------------|--------------------------|------|
| | <del></del> | |
| Name of Participant | Signature of Participant | Date |

# **Upholding Informed Consent Principles**

As the researcher, I am committed to upholding the highest ethical standards in ensuring informed consent. All questions the patient raised concerning the study and their potential involvement have been addressed truthfully and transparently. Furthermore, we have reaffirmed the voluntary nature of their participation, safeguarding their right to make an independent decision free from coercion or undue influence.

| safeguarding their right to make ar influence. | n independent decision free from | coercion or undue |
|---|---|---|
| By prioritizing transparency and re-<br>ethical principles that guide respon | | ain grounded in the |
| Signature of Researcher Who | Received Consent | |
| Name of Investigator | Signature of Investigator | Date |